CLINICAL TRIAL: NCT04902820
Title: PrEPTECH Phase 2 Study: Randomized-Controlled Trial of a Telehealth Intervention Delivering PrEP to Young Men Who Have Sex With Men and Transgender Women
Brief Title: PrEPTECH Phase 2 Study of a PrEP Telehealth Intervention
Acronym: PrEPTECH2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ETR Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PrEPTECH2
Record Dates: First submitted 2021-04-14; First posted 2021-05-26 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Pre-Exposure Prophylaxis; HIV; Telemedicine
Keywords: Randomized Controlled Trial; Online systems; Sexual and Gender Minorities; Transgender Persons; Adolescent; Sexual health
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Intervention Model Description: This is a two-arm randomized controlled trial with a one-to-one allocation ratio. Randomization will be stratified by sub-group (adult men who have sex with men ages 18-27 [n = 320], adult transgender women ages 18-27 [n = 40], and adolescent men who have sex with men ages 15-17 [n = 40]).
Masking Description: Participants are randomly assigned and will be made aware of the condition to which they are assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PrEPTECH intervention recipients (Experimental): The intervention is a web site delivering access to PrEP telehealth. The platform provides access to laboratory testing for PrEP eligibility delivered to a participant's home, telehealth care and PrEP prescriptions for those eligible delivered asynchronously through an online form for all adult participants and through telephone appointments for adolescent participants, and a mail-order pharmacy for PrEP. Additionally, free PrEP medication will be provided through the intervention. Transgender female and adolescent cisgender male participants will receive free PrEP medication (emtricitabine [200 mg]/tenofovir disoproxil fumarate [300 mg]) for the duration of their participation in the study, while adult cisgender male participants will receive a free 30-day supply of PrEP and subsequently have to pay for PrEP medication through insurance, patient assistance programs, or out of pocket.
  Interventions: Other: PrEPTECH website
- Control resource-list only recipients (Active Comparator): Participants will receive access to an online list of web-based resources about PrEP and how to locate and pay for PrEP care and contact information for a professional PrEP navigator at a local community-based organization partnering with the study.
  Interventions: Other: Online PrEP resource list

INTERVENTIONS:
Other: PrEPTECH website — The intervention is a web site delivering access to PrEP telehealth. The platform provides access to laboratory testing for PrEP eligibility delivered to a participant's home, telehealth care and PrEP prescriptions for those eligible delivered asynchronously through an online form for all adult participants and through telephone appointments for adolescent participants, and a mail-order pharmacy for PrEP. Additionally, free PrEP medication will be provided through the intervention. Transgender female and adolescent cisgender male participants will receive free PrEP medication (emtricitabine [200 mg]/tenofovir disoproxil fumarate [300 mg]) for the duration of their participation in the study, while adult cisgender male participants will receive a free 30-day supply of PrEP and subsequently have to pay for PrEP medication through insurance, patient assistance programs, or out of pocket.
  Arms: PrEPTECH intervention recipients
Other: Online PrEP resource list — Participants will receive access to an online list of web-based resources about PrEP and how to locate and pay for PrEP care and contact information for a professional PrEP navigator at a local community-based organization partnering with the study.
  Arms: Control resource-list only recipients

SUMMARY:
PrEPTECH Phase 2 is a 2-arm randomized controlled trial to assess the effectiveness of a telehealth intervention in increasing PrEP uptake among cisgender men and transgender women who have sex with men over six months. Participants (N = 400) will be randomized equally into one of two study conditions, treatment with a telehealth intervention called PrEPTECH or a control condition consisting of treatment as usual plus access to a listing of online and local PrEP resources, and assessed via surveys at baseline and at 90 and 180 days after baseline. Randomization of participants will be stratified by participant sub-group (adult men who have sex with men, adolescent men who have sex with men, and transgender women).

The baseline and follow-up assessments will include questions on demographic characteristics, measures related to our primary and secondary outcomes, and psychosocial measures. The primary outcomes measure is self-reported PrEP initiation at 3-month post enrollment, the percentage of participants reporting having taken at least one dose of PrEP medication by that time point. In addition, usage data and medical data will be collected and analyzed.

DETAILED DESCRIPTION:
A 2-arm randomized controlled trial will be conducted to assess the effectiveness of a telehealth intervention in increasing PrEP uptake among cisgender gay or bisexual men and transgender women over six months. PrEPTECH 2 is a follow-up to a pilot study of PrEPTECH undertaken in 25 adult men who have sex with men aged 18-25 years from the San Francisco Bay Area. In the pilot, PrEPTECH reached underserved populations, providing access to a pre-exposure prophylaxis (PrEP) regimen through a convenient telehealth system. The digital PrEPTECH 1 program provided digital PrEP education and resources to users, facilitated PrEP initiation and maintenance, simplified appointments needed to begin and maintain PrEP regimens through telemedicine appointments with physicians, eliminated the need for direct in-person follow-up with medical providers, provided a gay and bisexual male preferred telehealth method for accessing PrEP, offered personalized messaging to increase adherence and motivation for PrEP regimens, bypassed stigma and cost barriers for PrEP uptake in young men who have sex with men, and decreased the time required of clinicians managing PrEP patients. This follow-up study will extend our understanding of the PrEPTECH intervention and its capacity to increase PrEP uptake, adherence and maintenance, extending the populations served to include adolescent MSM ages 15-17 and transgender women.

In this phase 2 study, participants (N = 400) will be randomized equally into one of two study conditions, treatment with the PrEPTECH telehealth intervention or a control condition. Randomization of participants will be stratified by participant sub-group (adult men who have sex with men, adolescent men who have sex with men, and transgender women). Those in the treatment arm will have access to PrEPTECH for six months. PrEPTECH features includes a platform for connecting the participant with a prescribing physician providing free PrEP care, optional email or text message reminders, free home lab testing, and a supply of free PrEP (a 6 month supply for adolescent and transgender gender women participants and a 1 month supply for all other participants). Those in the control arm will be provided with a list of online resources about PrEP and how to locate and pay for PrEP care and contact information for a professional PrEP navigator at a local community-based organization partnering with the study. Participants will complete brief online surveys at baseline and at 90- and 180-days following baseline.

Participants will be recruited using a variety of methods, including through digital advertising on social media platforms and online dating/hook-up web sites and posting to community listservs, web sites offering resources on finding PrEP, and forums; community-based organizations partnering, that will assist with recruitment through social media and other online communication and in-person advertising with palm cards and flyers.

Randomization. Stratified randomization will be used to allocate participants. Participants will be stratified by study site and participant sub-group, ensuring that half of participants in each study site will be allocated to the PrEPTECH condition and half to the control condition and that the participants in each of the three study populations (adult YMSM, minors, and transgender women) will also be allocated equally to each of the two conditions.

Implementation. After randomization participants in the treatment group, will be granted access to the online PrEPTECH intervention, which includes a panel that sets-up text-message or email medication reminders, information about the intervention and PrEP, and a panel that guides the participant through the process of getting on PrEP: from ordering home lab testing, to completing a telehealth appointment with a study doctor, to ordering PrEP medication home delivery through an online pharmacy. Those in the control group will exclusively have access to a static web page offering links to online resources and information about local PrEP navigation resources available to them.

Data Collection. Participants will be surveyed at three time points: 1) prior to randomization (baseline) 2) 3 months (90 days) after enrollment 4) and 6 months (180 days) after enrollment. Surveys will be created on Qualtrics, hosted on the PrEPTECH web site, and taken online. All survey data will be transferred to SPSS for survey analysis. Data will also be collected through the app on usage of the web site. Additional study data will come from the lab tests collected prior to the first prescription being administered (hepatitis B, HIV, creatinine, serum creatinine and syphilis, gonorrhea, and chlamydia test) and roughly 90 days later (HIV, syphilis, gonorrhea and chlamydia).

ELIGIBILITY:
Inclusion Criteria:

* Live in the San Francisco Bay Area, CA (the 9-counties of Alameda, Contra Costa, Marin, Napa, San Mateo, Santa Clara, Solano, Sonoma, and San Francisco); Los Angeles County, CA; Miami-Dade County, FL; or Broward County, FL.
* Qualify for PrEP by virtue of self-reporting being diagnosed with a sexually transmitted infection (including chlamydia, genital herpes, gonorrhea, syphilis, genital warts, HPV, trichomoniasis, and other less common STIs) in the past six months or self-reporting unprotected anal intercourse in the past 90 days.
* Report having sex with men
* Either: Identify as a cisgender male and age 15-17 (in California only; minors in Broward or Miami-Dade Counties will not be eligible) OR identify as a cisgender male and age 18-27 OR identify as a transgender woman (or assigned male at birth and identify as a woman) and age 18-27

Exclusion Criteria:

* Must not have taken PrEP in the past 30 days
* Ever been diagnosed with HIV, hepatitis B, kidney disease, liver disease, or bone disease.
* Not meeting inclusion criteria

Ages: 15 Years to 27 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Transgender women and cis gender men are eligible.
Enrollment: 229 (Actual)
Dates: Start 2022-02-12 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Self-reported PrEP initiation | 3 months post enrollment
  Percentage of participants reporting having taken at least one dose of PrEP medication at any point during the intervention period

SECONDARY OUTCOMES:
Self-reported PrEP initiation | 6 months post enrollment
  Percentage of participants reporting having taken at least one dose of PrEP medication at any point during the intervention period
Self-reported PrEP persistence | 3 months post enrollment and 6 months post enrollment
  Percentage of participants reporting having taken at least one dose of PrEP medication during both the first and second 90-day periods of the intervention.
Self-reported PrEP adherence, continuous (3 months) | 3 months post enrollment
  Excluding participants taking event-based PrEP, the count of doses of PrEP taken in the past 30 days.
Self-reported PrEP adherence, continuous (6 months) | 6 months post enrollment
  Excluding participants taking event-based PrEP, the count of doses of PrEP taken in the past 30 days.
Self-reported PrEP adherence, categorical (3 months) | 3 months
  Excluding participants taking event-based PrEP, the percentage of participants who reported taking a dose of PrEP medication at least 4 days per week "All of the last 4 weeks (4 out of 4 weeks)" or "Most of the last 4 weeks (3 out of 4 weeks)"
Self-reported PrEP adherence, categorical (6 months) | 6 months
  Excluding participants taking event-based PrEP, the percentage of participants who reported taking a dose of PrEP medication at least 4 days per week "All of the last 4 weeks (4 out of 4 weeks)" or "Most of the last 4 weeks (3 out of 4 weeks)"
PrEP coverage at 3 months post-enrollment | 3 months post enrollment
  Number of instances of vaginal or anal sex in which there was no protection from event-driven PrEP (defined as taking PrEP between 2 and 24 hours ahead of the sex act(s) and 2 more doses 24 and 48 hours after the first dose) or continuous PrEP (defined as taking a minimum of 4 doses of PrEP within a week of the sex act(s)), past 30 days
PrEP coverage at 6 months post-enrollment | 6 months post enrollment
  Number of instances of vaginal or anal sex in which there was no protection from event-driven PrEP (defined as taking PrEP between 2 and 24 hours ahead of the sex act(s) and 2 more doses 24 and 48 hours after the first dose) or continuous PrEP (defined as taking a minimum of 4 doses of PrEP within a week of the sex act(s)), past 30 days
Self-reported PrEP medication prescription, self-reported | 3-months post enrollment and 6 months post enrollment
  Percentage of participants reporting having received a PrEP prescription at any point during the intervention period
PrEP medication prescription, observed | 3-months post enrollment and 6 months post enrollment
  Based on study records, percentage of participants who were issued a PrEP prescription through the study electronic health record at any point during the study period, amongst eligible intervention arm participants
System Usability Scale | 6 months post enrollment
  Among intervention arm participants, score on the scale ranging from 0 to 40, the sum of scores on 10 items, with higher scores indicating better usability, a better outcome.
Reported likelihood of recommending PrEPTECH | 6 months post enrollment
  Among intervention arm participants, percentage of participants reporting they "definitely" or "probably" would recommend PrEPTECH to a friend who wanted to start PrEP.
Reported interest in continuing in PrEPTECH beyond the study period | 6 months post enrollment
  Among intervention arm participants, percentage of participants who would "definitely" or "probably" want to continue using PrEPTECH if given the chance to at the end of the intervention.
Transition to community care | 6 months post enrollment
  Percentage of participants who are in the control group or opt to transition to community PrEP care during the course of the intervention who received a PrEP prescription in the past 90 days at 6-month post-enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Braun, DrPH, MPH, Principal Investigator — ETR
Locations (1):
- ETR, Scotts Valley, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Refugio ON, Kimble MM, Silva CL, Lykens JE, Bannister C, Klausner JD. Brief Report: PrEPTECH: A Telehealth-Based Initiation Program for HIV Pre-exposure Prophylaxis in Young Men of Color Who Have Sex With Men. A Pilot Study of Feasibility. J Acquir Immune Defic Syndr. 2019 Jan 1;80(1):40-45. doi: 10.1097/QAI.0000000000001873. PMID 30272632
- [Derived] Erenrich RK, Braun RA, Torres-Mendoza DM, Stevenson OL, Doan TP, Klausner JD. Effectiveness of PrEPTECH: Findings From a 180-Day Randomized Controlled Trial of a Pre-Exposure Prophylaxis Telehealth Intervention. J Acquir Immune Defic Syndr. 2024 Apr 15;95(5):463-469. doi: 10.1097/QAI.0000000000003375. Epub 2024 Mar 11. PMID 38133600
- [Derived] Braun RA, Erenrich RK, Coyle KK, Doan TP, Klausner JD. Effectiveness, Acceptability, and Feasibility of a Telehealth HIV Pre-Exposure Prophylaxis Care Intervention Among Young Cisgender Men and Transgender Women Who Have Sex With Men: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Sep 15;12:e47932. doi: 10.2196/47932. PMID 37713244